CLINICAL TRIAL: NCT00895947
Title: Evaluation of Natural Human Interferon Alpha Lozenges in the Prevention of Winter Colds and Flu in Perth, Western Australia
Brief Title: Interferon Alpha Lozenges in the Prevention of Winter Colds and Flu
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Collaborators: Department of Health, Western Australia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-113
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Prophylaxis; Treatment; Symptoms; Winter Colds and Flu
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human | interventions — Interferon-alpha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon-alpha (Experimental): 150 international units of interferon-alpha
  Interventions: Drug: interferon-alpha
- placebo (Placebo Comparator): placebo lozenges
  Interventions: Other: placebo

INTERVENTIONS:
Drug: interferon-alpha — a lozenge for oral dissolution containing 150 international units of human interferon-alpha taken once daily for 16 weeks
  Other Names: IFN-alpha lozenge
  Arms: Interferon-alpha
Other: placebo — placebo lozenges for oral dissolution taken once daily for 16 weeks
  Other Names: Maltose lozenge
  Arms: placebo

SUMMARY:
The aim of the study is to see if lozenges containing a low dose of interferon-alpha can prevent and/or reduce the severity of colds and flu. Starting about 1 month before the expected start of the winter colds and flu season in Perth, Australia, healthy volunteers will allow a lozenge containing interferon, or a lozenge containing no medicine (a placebo), to dissolve in their mouth once a day for 16 weeks. Blood tests at the start and end of treatment will determine whether interferon was able to prevent infections with cold/flu viruses. Once a week, volunteers will complete a survey about their cold/flu symptoms, medications taken, days of work missed, etc. to see if interferon was able to make their winter colds and flu less severe.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* Females of child-bearing potential must practice a medically accepted form of birth control

Exclusion Criteria:

* Currently exhibiting an acute upper respiratory tract infection
* history of chronic respiratory disease requiring regular therapy(i.e. COPD, asthma, bronchitis, etc.)
* any condition likely to increase the risk of severe or complicated influenza (i.e. cardiac disease, chronic renal disease, endocrine diseases, including diabetes and/or immunosuppressive therapy)
* any condition requiring regular treatment with antihistamines, analgesics or antipyretics
* known infection with HIV, hepatitis B virus or hepatitis C virus
* any other serious, uncontrolled disease
* any active infections requiring use of antibiotic or antiviral drugs
* non-ambulatory status
* suspected drug or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, PhD, Principal Investigator — Path West Laboratory Medicine WA
Locations (1):
- University of Western Australia, Nedlands, Western Australia, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 healthy volunteers were enrolled at the University of Western Australia in Perth between April 17 and July 31, 2009.
Pre-assignment Details: Two of 200 randomized subjects (one in each group) decided not to begin study treatment after enrollment, so only 198 subjects were evaluable for response.
Groups:
- Interferon-alpha: 150 international units of interferon-alpha given once daily for 16 weeks in an orally disolving lozenge consisting of 200 mg of anhydrous crystalline maltose
- Placebo: 200 mg anhydrous crystalline maltose given once daily for 16 weeks in an orally disolving lozenge
Period: Overall Study
Arm/Group | Interferon-alpha | Placebo
Started | 100 | 100
Completed | 88 | 90
Not Completed | 12 | 10
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon-alpha | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 91 | 186
  >=65 years | 5 | 9 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (14.4) | 47.3 (13.2) | 46.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 66 | 136
  Male | 30 | 34 | 64
Region of Enrollment [Number; unit: participants]
  Australia | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Influenza-like Illness
Description: Number of subjects in each group meeting the definition of influenza-like illness during treatment (i.e. those subject reporting one or more moderate to severe cold/flu symptoms during the treatment period).
Time Frame: 16 weeks
Population: Intent-to-treat, defined as all randomized subjects who took at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  Overall | 54 | 62
  Age 50 and over | 16 | 28
  Age under 50 | 38 | 34
  Seasonal flu vaccine, yes | 16 | 36
  Seasonal flu vaccine, no | 38 | 26
  Gender, Male | 11 | 22
  Gender, Female | 43 | 40
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.25, Chi-squared — Overall comparison of treatment groups for incidence of ILI
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.01, Chi-squared — Comparision of ILI incidence in subjects age 50 and older at baseline
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.32, Chi-squared — Comparison of ILI in subjects age < 50 at baseline
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.01, Chi-squared — Comparison of ILI incidence in subjects vaccinated against seasonal influenza prior to enrollment
Statistical Analysis 5: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.45, Chi-squared — Comparison of ILI incidence in subjects not vaccinated against seasonal influenza prior to enrollment
Statistical Analysis 6: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared — Comparison of ILI incidence in male subjects
Statistical Analysis 7: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.99, Chi-squared — Comparison of ILI incidence in female subjects

2. Secondary Outcome: Symptom Incidence/Severity
Description: Number of subjects in each group reporting 13 different cold/flu symptoms assessed weekly
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  any cold/flu symptoms | 86 | 92
  moderate to severe feverishness | 12 | 24
  moderate to severe head congestion | 23 | 36
  moderate to severe sore throat | 27 | 39
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.16, Chi-squared — Proportion of subjects reporting any cold/flu symptoms during treatment
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared — Proportion of subjects reporting moderate to severe feverishness
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.04, Chi-squared — Proportion of subjects reporting moderate to severe head congestion
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.07, Chi-squared — Proportion of subjects reporting moderate to severe sore throat

3. Secondary Outcome: Impact of Cold/Flu Symptoms
Description: Number of subjects in each group reporting that cold/flu symptoms impacted the following 9 measures of daily life: ability to (1) think clearly, (2) sleep well, (3) breathe easily, (4) walk, climb stairs and exercise, (5) perform daily tasks, (6) work outside the home, (7) work inside the home, (8) interact with others, and (9) live personal life.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  think clearly | 53 | 59
  sleep well | 54 | 64
  breathe easily | 58 | 61
  walk, climb stairs and exercise | 44 | 49
  perform daily activities | 46 | 54
  work outside the home | 43 | 51
  work inside the home | 42 | 51
  interact with others | 41 | 50
  live personal life | 44 | 51
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.39, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to think clearly
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.15, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to sleep well
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.66, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to breathe easily
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.48, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to walk, climb stairs and exercise
Statistical Analysis 5: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.26, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to perform daily activities
Statistical Analysis 6: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.25, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to work outside the home
Statistical Analysis 7: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.20, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to work inside the home
Statistical Analysis 8: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.20, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to interact with others
Statistical Analysis 9: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.32, Chi-squared — Proportion of subjects reporting one of more days that cold/flu symptoms impacted ability to live personal life

4. Secondary Outcome: Negative Events Related to Cold/Flu Symptoms
Description: Number of subjects in each group reporting one or days of occurrence of the following 6 negative events: (1) felt sick, (2) missed work, (3) went to the doctor, (4) went to the pharmacy, (5) took cold/flu medication, and (6) skipped a planned activity
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  felt sick | 62 | 65
  missed work | 32 | 33
  visited the doctor | 16 | 16
  visited the pharmacy | 34 | 30
  took cold/flu medication | 57 | 65
  skipped a planned activity | 46 | 45
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.66, Chi-squared — Proportion of subjects in each group reporting one or more days they felt sick
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.88, Chi-squared — Proportion of subjects in each group reporting one or more days they missed work
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 1.0, Chi-squared — Proportion of subjects in each group reporting one or more days they visited the doctor
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.54, Chi-squared — Proportion of subjects in each group reporting one or more days they visited the pharmacy
Statistical Analysis 5: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.24, Chi-squared — Proportion of subjects in each group reporting one or more days they took cold/flu medication
Statistical Analysis 6: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.89, Chi-squared — Proportion of subjects in each group reporting one or more days they skipped a planned activity

5. Secondary Outcome: Incidence/Severity of Viral Respiratory Infections
Description: Number of subjects in each group with a confirmed viral respiratory infection and the proportion of subjects reporting a mild vs. moderate to severe infection
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  incidence of viral respiratory infection | 20 | 23
  moderate/severe viral respiratory infection | 5 | 16
  moderate/severe influenza infection | 1 | 4
  moderate/severe non-influenza infection | 4 | 11
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.61, Chi-squared — Proportion of subjects in each group with a confirmed viral respiratory infection
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.003, Chi-squared — Proportion of subjects in each group with a moderate/severe viral respiratory infection
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared — Proportion of subjects in each group with a moderate/severe influenza infection
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared — Proportion of subjects in each group with a moderate/severe viral respiratory infection other than influenza

6. Post Hoc Outcome: Acute Respiratory Illness
Description: Number of subjects in each group meeting definition of acute respiratory illness (ARI), defined as 2 or more cold/flu symptoms reported in the same week. Further defined as "febrile" or "afebrile" depending on whether the subject reported the symptom of "feverishness."
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Interferon-alpha | Placebo
Number analyzed (Participants) | 99 | 99
participants
  all acute respiratory illness (ARI) | 83 | 86
  moderate/severe ARI | 41 | 54
  moderate/severe febrile ARI | 12 | 24
  moderate/severe afebrile ARI | 35 | 31
Statistical Analysis 1: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.54, Chi-squared — Proportion of subjects meeting the definition of acute respiratory illness during treatment
Statistical Analysis 2: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.06, Chi-squared — Proportion of subjects meeting with moderate/severe acute respiratory illness during treatment
Statistical Analysis 3: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.03, Chi-squared — Proportion of subjects with moderate/severe febrile acute respiratory illness during treatment
Statistical Analysis 4: Comparison: Interferon-alpha vs Placebo; Test type: Superiority or Other; p = 0.60, Chi-squared — Proportion of subjects with moderate/severe afebrile acute respiratory illness during treatment

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Interferon-alpha | Placebo
Serious Adverse Events (participants affected / at risk) | 1/99 | 1/99
Other Adverse Events (participants affected / at risk) | 30/99 | 33/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon-alpha (N=99) | Placebo (N=99)
appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — subject underwent an emergency appendectomy judged by the attending investigator to be unrelated to study medication
hemorroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — subject underwent an emergency hemorroidectomy judged by the attending investigator to be unrelated to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon-alpha (N=99) | Placebo (N=99)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8)
diarrhea (Gastrointestinal disorders) | 14 (20) | 9 (12)
fatigue (General disorders) | 4 (5) | 8 (9)
hay fever (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 13 (17)
headache (Nervous system disorders) | 11 (20) | 10 (14)
migraine (Nervous system disorders) | 4 (4) | 5 (10)
nausea (Gastrointestinal disorders) | 5 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No